CLINICAL TRIAL: NCT01774812
Title: Vitamin D Supplementation and Cardiac Autonomic Tone in Hemodialysis Patients: A Blinded, Randomized-controlled Trial
Brief Title: Vitamin D and Cardiac Autonomic Tone in Hemodialysis
Acronym: VITAH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Sofia Ahmed, Dr. Sofia B. Ahmed, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UC-Neph-2012001
Record Dates: First submitted 2013-01-17; First posted 2013-01-24 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Cardiovascular Disease; Sudden Cardiac Death
Keywords: vitamin D; hemodialysis; sudden cardiac death; heart rate variability; cardiac autonomic tone
MeSH Terms: conditions — Cardiovascular Diseases; Death, Sudden, Cardiac | interventions — alfacalcidol; Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D Sequence 1 (Active Comparator): 6 weeks - alfacalcidol 0.25mcg + placebo 3x per week, 12 week washout, 6 weeks - alfacalcidol 0.25mcg 3x per week + 50,000IU ergocalciferol 1x per week (placebo the 2 remaining days)
  Interventions: Dietary Supplement: Alfacalcidol; Dietary Supplement: Ergocalciferol
- Vitamin D Treatment Sequence 2 (Active Comparator): 6 weeks - alfacalcidol 0.25mcg 3x per week + 50,000IU ergocalciferol 1x per week (placebo the 2 remaining days), 12 week washout, 6 weeks - alfacalcidol 0.25mcg + placebo 3x per week
  Interventions: Dietary Supplement: Alfacalcidol; Dietary Supplement: Ergocalciferol

INTERVENTIONS:
Dietary Supplement: Alfacalcidol — 0.25 mcg 3x per week for 6 weeks
Dietary Supplement: Ergocalciferol — 50,000IU 1x per week for 6 weeks

SUMMARY:
Despite advances in treatment of conventional cardiovascular risk factors, patients with kidney disease remain at high risk for fatal cardiac events. To date, kidney disease affects approximately 2 million Canadians; however, this patient population remains grossly understudied due to the complex nature of the disease. The inadequacy of the literature to address the cardiovascular-related mortality rates in those with kidney disease reflects the urgent need for investigation of novel risk factors.

One cardiovascular risk factor which has recently been validated is the clinical measurement of cardiac autonomic tone (CAT). CAT refers to the amount of activity contributed by the stimulatory and inhibitory limbs of the cardiac autonomic nervous system, which work in concert with one another to control heart rate. CAT can be quantified computer analysis of heart rate over time, captured by a simple Holter electrocardiogram (ECG) recording. Abnormal CAT, which occurs when the autonomic system does not control heart rate properly in response to physical demands or stress, is associated with risk of adverse cardiovascular events in both healthy and high risk populations. It has recently been shown that patients with severe kidney disease demonstrate significant CAT abnormalities, thus exaggerated susceptibility to cardiac death.

Vitamin D (VD) deficiency is also common in this patient population due to the fact that the kidney plays a crucial role in VD metabolism. Given that VD deficiency is an established cardiovascular risk factor on its own, it is possible that kidney disease patients experienced compounded risk due to the combination of VD deficiency and abnormal CAT. However, no study has ever investigated whether VD deficiency influences CAT in healthy or diseased populations. To our knowledge, this will be the first trial to ever examine the effect, if any, of different VD supplementation treatments (standard of care vs. combination) on CAT in a population burdened with overwhelming risk and incidence of cardiovascular and sudden cardiac death risk.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* 3x weekly hemodialysis outpatient within Calgary for at least 3 months prior to enrolment
* physician consent to participate in VD supplementation regimen
* ability and agreement to cease any VD medication for 4 weeks prior to initiation of study
* able to comprehend study and provide oral and written consent in English

Exclusion Criteria:

* any major cardiovascular event (new onset arrhythmia, hospitalization for a cardiac event) noted in patient chart within the 6 month period prior to initiation of the study
* currently on VD therapy/refusal to cease VD therapy for 4 weeks prior to initiation of study
* physician anticipates death or adverse event within the next year- known discharge from hemodialysis (transfer to peritoneal dialysis, kidney transplant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
LF:HF | change from baseline to 6 weeks
  Low frequency to high frequency ratio (sympathetic vs. parasympathetic cardiac autonomic power)
LF:HF | change from 6 weeks to 18 weeks
  Low frequency to high frequency ratio (sympathetic vs. parasympathetic cardiac autonomic power)
LF:HF | change from 18 weeks to 24 weeks
  Low frequency to high frequency ratio (sympathetic vs. parasympathetic cardiac autonomic power)

SECONDARY OUTCOMES:
SDNN | every 6 weeks up to 24 weeks
  standard deviation of normal wave (heart rate variability time domain)
SDANN | every 6 weeks up to 24 weeks
  standard deviation of the average normal wave (heart rate variability time domain)
pNN50% | every 6 weeks up to 24 weeks
  percentage of normal waves which differ in frequency > 50 ms compared to the wave directly before (heart rate variability time domain)
LF | every 6 weeks up to 24 weeks
  Low-frequency (ms squared and normalized units), thought to reflect sympathetic contribution from the cardiac autonomic nervous system
HF | every 6 weeks up to 24 weeks
  High-frequency (ms squared and normalized units), thought to reflect parasympathetic contribution from the cardiac autonomic nervous system

OTHER OUTCOMES:
25-hydroxy vitamin D | every 6 weeks up to 24 weeks
1,25-dihydroxyvitamin D | every 6 weeks up to 24 weeks
Parathyroid hormone | every 6 weeks up to 24 weeks
Calcium | every 6 weeks up to 24 weeks
Phosphate | every 6 weeks up to 24 weeks
Pre- and post-dialysis weight | every 6 weeks up to 24 weeks
Epinephrine | every 6 weeks up to 24 weeks
Norepinephrine | every 6 weeks up to 24 weeks
Renin-angiotensin system activity (circulating) | every 6 weeks up to 24 weeks
  renin, angiotensin II, aldosterone

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sofia B Ahmed, MD, MMSc, Principal Investigator — University of Calgary; Dr. Derek Exner, MD, MPH, Principal Investigator — University of Calgary, Libin Cardiovascular Institute; Dr. Brenda Hemmelgarn, MD, PhD, MN, Principal Investigator — University of Calgary
Locations (3):
- Canada (3):
  - Northland Hemodialysis Clinic, Calgary, Alberta
  - Foothills Medical Centre - University of Calgary, Calgary, Alberta
  - Sheldon M. Chumir Health Centre, Calgary, Alberta

REFERENCES:
- [Background] Mann MC, Exner DV, Hemmelgarn BR, Turin TC, Sola DY, Ahmed SB. Impact of gender on the cardiac autonomic response to angiotensin II in healthy humans. J Appl Physiol (1985). 2012 Mar;112(6):1001-7. doi: 10.1152/japplphysiol.01207.2011. Epub 2012 Jan 5. PMID 22223455
- [Background] Drechsler C, Pilz S, Obermayer-Pietsch B, Verduijn M, Tomaschitz A, Krane V, Espe K, Dekker F, Brandenburg V, Marz W, Ritz E, Wanner C. Vitamin D deficiency is associated with sudden cardiac death, combined cardiovascular events, and mortality in haemodialysis patients. Eur Heart J. 2010 Sep;31(18):2253-61. doi: 10.1093/eurheartj/ehq246. Epub 2010 Aug 5. PMID 20688781
- [Background] Lahiri MK, Kannankeril PJ, Goldberger JJ. Assessment of autonomic function in cardiovascular disease: physiological basis and prognostic implications. J Am Coll Cardiol. 2008 May 6;51(18):1725-33. doi: 10.1016/j.jacc.2008.01.038. PMID 18452777
- [Background] Mann MC, Exner DV, Hemmelgarn BR, Sola DY, Turin TC, Ellis L, Ahmed SB. Vitamin D levels are associated with cardiac autonomic activity in healthy humans. Nutrients. 2013 Jun 10;5(6):2114-27. doi: 10.3390/nu5062114. PMID 23752493
- [Derived] Mann MC, Exner DV, Hemmelgarn BR, Hanley DA, Turin TC, MacRae JM, Wheeler DC, Sola DY, Ramesh S, Ahmed SB. The VITAH Trial-Vitamin D Supplementation and Cardiac Autonomic Tone in Patients with End-Stage Kidney Disease on Hemodialysis: A Blinded, Randomized Controlled Trial. Nutrients. 2016 Sep 28;8(10):608. doi: 10.3390/nu8100608. PMID 27690095
- [Derived] Mann MC, Exner DV, Hemmelgarn BR, Hanley DA, Turin TC, MacRae JM, Ahmed SB. The VITAH trial VITamin D supplementation and cardiac Autonomic tone in Hemodialysis: a blinded, randomized controlled trial. BMC Nephrol. 2014 Aug 6;15:129. doi: 10.1186/1471-2369-15-129. PMID 25098377